CLINICAL TRIAL: NCT02708628
Title: The Efficacy of Prophylactic Use of Extract of Allium Cepae, Allantoin and Heparin in Patients With Proven Scar Development After Excision of Previous Scar
Brief Title: The Efficacy of Extract of Allium Cepae, Allantoin and Heparin in Patients With Proven Scar Development
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suleymaniye Birth And Women's Health Education And Research Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AGZ-EAC-A-H-1
Record Dates: First submitted 2016-02-29; First posted 2016-03-15 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-03

CONDITIONS: Cicatrix
Keywords: scar prevention; sectio; extract of allium cepae; allantoin; heparin
MeSH Terms: conditions — Cicatrix | interventions — Allantoin; Heparin; allantoin, heparin, onion extract drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients using contractubex (Active Comparator): Scar excision will be performed in second c-section for 60 patients and these patients will use prophylactic topical scar gel containing extract of allium cepae, allantoin and heparin two times in a day.
  Interventions: Drug: extract of allium cepae, allantoin and heparin; Procedure: Scar excision
- Patients not using contractubex (Active Comparator): Scar excision will be performed in second c-section for 60 patients and these patients will not use prophylactic topical scar gel containing extract of allium cepae, allantoin and heparin.
  Interventions: Procedure: Scar excision

INTERVENTIONS:
Drug: extract of allium cepae, allantoin and heparin — prophylactic use of a topical gel containing extract of allium cepae, allantoin and heparin two times in a day after second c-section
  Other Names: Contractubex
  Arms: Patients using contractubex
Procedure: Scar excision — Scar excision in second c-section

SUMMARY:
To investigate the efficacy of prophylactic use of a topical gel containing extract of allium cepae, allantoin and heparin after surgical removal of the primary cesarean scar in the second cesarean section.

DETAILED DESCRIPTION:
120 patients who are admitted for the second cesarean delivery, not taking prophylactic medication after the first cesarean section, whose scar development and measurements are taken will be included in the study. First caesarean section scars will be removed surgically for all patients. 60 out of 120 patients (treatment group) will use prophylactic topical scar gel 2 times in a day, and remaining 60 patients (control group )won't use. The efficacy of the drug will be evaluated by taking strict measurements of the incision and POSAS (The Patient and Observer Scar Assessment Scale) and Vancouver Scales at 6.12 and 24 weeks.

Steps;

1. Observation of the primary cesarean scar by taking scar measurements and using Vancouver and POSAS scales.
2. Surgical removal of the primary cesarean scar in the second cesarean section.
3. 24 weeks topical application of gel containing extract of allium cepae, allantoin and heparin(only treatment group).
4. Observation of the skin incision at 6,12 and 24 weeks by taking scar measurements with using Vancouver and POSAS scales.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are admitted for the second cesarean delivery
* Not to use topical scar gel after the first c-section

Exclusion Criteria:

* chronic illness, immunosuppressive therapy or smoking
* development of wound infection during the second c- section
* allergies and hypersensitivities to components of the gel

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2015-12; Primary Completion 2016-04 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
POSAS observer score change will be assessed by POSAS observer scale (The Patient and Observer Scar Assessment Scale v2.0) just prior to second c-section and at 6,12 and 24 weeks following the c-section. | just prior to second c-section and at 6,12,24 weeks
POSAS patient score change will be assessed by POSAS patient scale (The Patient and Observer Scar Assessment Scale v2.0) just prior to second c-section and at 6,12 and 24 weeks following the c-section. | just prior to second c-section and at 6,12,24 weeks
Vancouver scar score change will be assessed by Vancouver scar scale just prior to second c-section and at 6,12 and 24 weeks following the c-section. | just prior to second c-section and at 6,12,24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ali Galip Zebitay, M.D., Principal Investigator — Suleymaniye Birth And Women's Health Education And Research Hospital
Locations (1):
- Suleymaniye Birth And Women's Health Education And Research Hospital., Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided